CLINICAL TRIAL: NCT01381809
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating Epoetin Alfa Versus Placebo in Anemic Patients With IPSS Low- or Intermediate-1-Risk Myelodysplastic Syndromes
Brief Title: An Efficacy Study for Epoetin Alfa in Anemic Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR018367; EPOANE3021 (Other: Janssen-Cilag International NV); 2010-022884-36 (EudraCT Number)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Myeloproliferative Disorders; Bone Marrow disease; Anemia; Epoetin Alfa; Eprex; Erypo; Erythropoiesis-stimulating agent
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Bone Marrow Diseases; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epoetin alfa (Experimental): Group 1: Epoetin alfa type = range unit= IU/Kg number= 337.5 to 1050 IU/Kg form= solution for injection route= subcutaneous use weekly injections (max 40 000 IU per week for first 8 weeks of treatment max 80 000 IU per week later) using pre-filled 1mL 40 000 IU syringes for 24 to 48 weeks
  Interventions: Drug: Group 1: Epoetin alfa
- No treatment (Placebo Comparator): Group 2: Placebo form= solution for injection route= subcutaneous use weekly injections for 24 to 48 weeks
  Interventions: Drug: Group 2: Placebo

INTERVENTIONS:
Drug: Group 2: Placebo — form= solution for injection, route= subcutaneous use, weekly injections for 24 to 48 weeks
  Arms: No treatment
Drug: Group 1: Epoetin alfa — type = range, unit= IU/Kg, number= 337.5 to 1050 IU/Kg, form= solution for injection, route= subcutaneous use, weekly injections (max 40,000 IU per week for first 8 weeks of treatment, max 80,000 IU per week later) using pre-filled 1mL 40,000 IU syringes for 24 to 48 weeks
  Arms: Epoetin alfa

SUMMARY:
The purpose of this study is to demonstrate that epoetin alfa works better than placebo in improving anemia in patients with lower-risk myelodysplastic syndromes (MDS). The safety of epoetin alfa will also be evaluated.

DETAILED DESCRIPTION:
This is a randomized (the treatment you receive will be assigned by chance), double-blind (neither physician nor patient knows the name of the assigned drug), placebo-controlled (comparison with patients that receive treatment without active ingredient), multicenter study of epoetin alfa in anemic patients who are diagnosed with myelodysplastic syndromes (MDS) according to protocol-specified criteria. This study includes a 3-week prerandomization phase, a 24-week treatment phase and a 24-week treatment extension phase. All patients enrolled in the study will complete an end-of-study visit 4 weeks after the last dose of study drug (Week 28 or Week 52), or 4 weeks after early withdrawal (unless the reason for early withdrawal is withdrawal of consent). Between 125 and 159 patients will be enrolled in the treatment phase of the study. During the screening phase, which will take place within 2 weeks before starting study drug, the study doctor will do tests to see if the patient is suitable for this study. Patients meeting entry criteria for the study will then be randomly assigned to one of the 2 treatment groups. This means that each patient who is allowed to join the study is put into a group by chance, like flipping a coin. Group 1 patients will receive epoetin alfa 450 or increased up to 1050 International Units (IU) per kg body weight administered by subcutaneous injection (injection beneath the skin) using pre-filled syringes. Injections will be done once every week at a weight-based dose regimen (the total weekly dose received will depend on your weight) with a possible total maximum dose of 40,000 IU once every week for the first 8 weeks of the treatment phase and 80,000 IU once every week at any other time during the study. Group 2 patients will receive a matching volume of placebo administered once every week by subcutaneous injection. The chance that the patient will get epoetin alfa is 2 to 1. Doses of study drug will be withheld, decreased, or increased on the basis of erythroid response, weekly hemoglobin concentrations monitored in patients and predefined dose adjustment guidelines. Patients will see the study doctor every 4 weeks for a period of 24 weeks. At each visit the patient will undergo a full hematologic evaluation, serum chemistry evaluation, measurement of blood pressure and pulse rate, recording of blood product transfusions and transfusion complications, adverse events, concomitant therapies and an evaluation for disease progression. The patient's Erythroid response will be assessed at Week 8 and every 4 weeks thereafter, until Week 24. Blinded study treatment will be administered to all patients at Week 24. However, at the end of the treatment phase (after the Week 24 response assessment), only responders will enter the double-blind treatment extension phase to measure the duration of response. Patients will continue to receive the same treatment, in the same blinded fashion, and at the same dose as received at Week 24, and will return to the study center every 4 weeks, until Week 48, for assessment of the Erythroid response and the evaluations as described above. For all non-responders at Week 24 the treatment code will be broken after Week 28 assessments. For responders at Week 48, the treatment code will be broken after the Week 48 visit, following completion of the response assessment. The treatment code will not be broken for subjects who discontinue study treatment before Week 24, irrespective of whether they are responders or nonresponders. For these subjects, the blind will not be broken until all subjects have completed the study and the database is final. Once the patient stops receiving doses of study drug, he/she will be asked to see the study doctor for the safety follow-up visit, which is scheduled 4 weeks after the last dose of study drug. Safety will be monitored throughout the study at predetermined intervals and as clinically indicated by physical examination, laboratory tests and evaluation of adverse events. An Independent Data Monitoring Committee (IDMC) will periodically review study data and for the assessment of disease progression. The total duration of study participation will be for about 30 or 54 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS according to World Health Organization or French-American-British pathologic classification (confirmed via bone marrow aspirate/biopsy) within 12 weeks prior to screening
* Documentation of an International Prognostic Scoring System score indicating Low- or Intermediate-1-risk disease within 12 weeks prior to screening
* Hemoglobin concentration at screening and baseline (before the first dose of study drug) of 10.0 g/dL or less
* Screening serum erythropoietin concentration of less than 500 mU/mL
* Red Blood Cell transfusion requirement of less than or equal to 4 red blood cell units over the last 8 weeks before randomization

Exclusion Criteria:

* Anemia attributed to factors other than MDS (including hemolysis, chronic renal failure, hepatitis, gastrointestinal bleeding)
* Secondary MDS (ie, MDS arising after chemotherapy, immunotherapy or radiation therapy/exposure)
* History of malignancy, except in situ skin basal cell carcinoma or carcinoma in situ of the cervix or breast curatively treated
* Prior therapy with any erythropoiesis-stimulating agent (ESA) (including innovative ESAs and biosimilar ESAs for approved indications or for investigational use) in the last 8 weeks before randomization
* Prior use of approved or experimental agents for the treatment of MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Erythroid response | at week 24

SECONDARY OUTCOMES:
Maintenance of Erythroid response | every 4 weeks from week 24 to week 48
Duration of response | every 4 weeks after week 24
Time to first Red Blood Cell transfusion | from baseline to study end (week 28 for non responders, week 54 for responders or 4 weeks after early withdrawal)
Transfusion-free intervals | from baseline to study end (week 28 for non responders, week 54 for responders or 4 weeks after early withdrawal)
Number of Red Blood Cell units transfused | from baseline to study end (week 28 for non responders, week 54 for responders or 4 weeks after early withdrawal)
Quality of life as measured by Functional Assessment of Cancer Therapy-Anemia/Fatigue (FACT-An) questionnaire | at baseline, week 24 and week 48
Quality of life as measured by EuroQol 5-dimension (EQ-5D) questionnaire | at baseline, week 24 and week 48
Drug consumption | every 4 weeks from baseline to week 48
Duration of hospitalization | every 4 weeks from baseline to week 48
Number and duration of medical care encounters | every 4 weeks from baseline to week 48

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (28):
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- France (10):
  - Amiens
  - Angers
  - Bobigny
  - Colmar
  - Paris
  - Pessac
  - Pierre-Bénite
  - Saint-Priest-en-Jarez
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (8):
  - Berlin
  - Dresden
  - Duisburg
  - Düsseldorf
  - Dÿsseldorf
  - München
  - Oldenburg
  - Würzburg
- Greece (5):
  - Athens
  - Goudi-Athens
  - Larissa
  - Pátrai
  - Thessalonikis
- Russia (2):
  - Saint Petersburg
  - Yekaterinburg

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating Epoetin Alfa Versus Placebo in Anemic Patients With IPSS Low- or Intermediate-1-Risk Myelodysplastic Syndromes — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=1105&filename=CR018367_CSR.pdf